CLINICAL TRIAL: NCT00003011
Title: A Phase III Study of Marimastat in Patients With Small Cell Lung Cancer Following a Response to First Line Chemotherapy
Brief Title: Marimastat Following Chemotherapy in Treating Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR12; EORTC-08962 (Other: EORTC); CAN-NCIC-BR12 (Registry Identifier: PDQ registration number); CDR0000065589 (Registry Identifier: PDQ registration number)
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — marimastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marmistat (Active Comparator): 10 mg PO BID
  Interventions: Drug: marimastat
- Placebo (Placebo Comparator): 10 mg PO BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: marimastat — 10 mg PO BID
  Arms: Marmistat
Drug: Placebo — 10 mg PO BID
  Arms: Placebo

SUMMARY:
RATIONALE: Marimastat may stop the growth of lung cancer by stopping blood flow to the tumor. It is not yet known if marimastat is an effective treatment for small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of marimastat with a placebo following chemotherapy in treating patients who have small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether treatment with the oral matrix metalloproteinase inhibitor (MMPI) marimastat prolongs overall survival and time to progression in patients with small cell lung cancer who have achieved complete or partial remission after first line chemotherapy, with or without radiotherapy. II. Determine the tolerability and toxicity of prolonged administration of marimastat in patients with small cell lung cancer. III. Determine the effect of prolonged administration of marimastat on the quality of life of patients with small cell lung cancer.

OUTLINE: This is a randomized, double blind, multicenter, placebo controlled study. Patients are stratified by stage of disease at diagnosis, response to prior chemotherapy/radiotherapy, type of thoracic radiotherapy, and cooperative group. Patients are randomized into two groups. Half of the patients take marimastat orally twice a day (breakfast and evening meal); the other half take placebo orally twice a day (breakfast and evening meal). Treatment continues for 2 years or until documented disease recurrence or progression and institution of further anticancer treatment, occurrence of unacceptable toxicity, initiation of anticoagulant treatment, or development of intercurrent illness. All patients are followed every 6 months until death.

PROJECTED ACCRUAL: The planned sample size is 360, with an equal number of patients in both arms, accrued at a rate of 240 responders per year (resulting in an accrual period of approximately 1.5 years). The total duration of the study is estimated as 2.3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven small cell lung cancer Complete response (CR) or partial response (PR) following first line chemotherapy required Chest x-ray showing CR or PR required. No documented prior brain metastases

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Effective contraception use by men or women of reproductive potential No prior malignancies within 5 years except: Adequately treated nonmelanomatous skin cancer Adequately treated carcinoma in situ of the cervix No other concurrent malignancies No prior diagnosis of breast cancer, melanoma, or hypernephroma No major medical illness that would preclude prolonged administration of marimastat or required follow up No active peptic ulceration or symptoms suggestive of this diagnosis No grade 3 or 4 musculoskeletal disorders

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: One prior induction combination chemotherapy regimen required Must be completed prior to randomization Hematologically recovered before randomization Minimum of 4 cycles required No change in regimen due to progression No chemotherapy within 28 days prior to randomization if thoracic radiation is given prior to or concurrent with chemotherapy No prior marimastat Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed Must be completed prior to randomization Last dose of radiation treatment must be within 7-14 days prior to randomization if thoracic radiation and/or prophylactic cranial irradiation is given after completion of chemotherapy If severe esophagitis precludes administration of oral medication, randomization may be within 21 days after radiation therapy Surgery: No surgery within 2 weeks prior to randomization Prior complete resection of tumor allowed Other: No other investigational agents within 4 weeks prior to study, and none planned No concurrent coumarin anticoagulants and no coumarin anticoagulants within 4 weeks prior to randomization No concurrent antitumor treatment

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 1997-01-31 (Actual); Primary Completion 2001-02-13 (Actual); Study Completion 2008-12-15 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 4 years
  To determine whether treatment with the oral metalloproteinase inhibitor marimastat prolongs overall survival and time to progression in patients with small cell lung cancer who have achieved complete or partial remission after first line chemotherapy (+I- radiotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD, PhD, Study Chair — Free University Medical Center; Frances A. Shepherd, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (38):
- Canada (38):
  - Cross Cancer Institute, Edmonton, Alberta
  - Penticton Regional Hospital, Penticton, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - York County Hospital, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huisman C, Postmus PE, Giaccone G, Smit EF. Second-line chemotherapy and its evaluation in small cell lung cancer. Cancer Treat Rev. 1999 Aug;25(4):199-206. doi: 10.1053/ctrv.1999.0125. PMID 10448128
- [Result] Shepherd FA, Giaccone G, Seymour L, Debruyne C, Bezjak A, Hirsh V, Smylie M, Rubin S, Martins H, Lamont A, Krzakowski M, Sadura A, Zee B. Prospective, randomized, double-blind, placebo-controlled trial of marimastat after response to first-line chemotherapy in patients with small-cell lung cancer: a trial of the National Cancer Institute of Canada-Clinical Trials Group and the European Organization for Research and Treatment of Cancer. J Clin Oncol. 2002 Nov 15;20(22):4434-9. doi: 10.1200/JCO.2002.02.108. PMID 12431965